CLINICAL TRIAL: NCT05470712
Title: A Retrospective Study of Vital Mechanism of NETs Formation vs. Suicidal Mechanism of NETs Formation During Normal Pregnancy and Preeclampsia
Brief Title: Vital Mechanism of NETs Formation vs. Suicidal Mechanism of NETs Formation During Normal Pregnancy and Preeclampsia
Acronym: GrossNETs
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2022-1/SB-01
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-02

CONDITIONS: Pre-Eclampsia
Keywords: Pregnancy; Pre-eclampsia; Neutrophils; Extracellular traps
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This study is based on the NETs formation mechanism of frozen plasma samples from patients included in a previous cohort (RCB 2014-A01120-47, NCT01736826). The benefits will ultimately be a better understanding of the physiopathological mechanisms involved in the occurrence of this placental vascular pathology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plasma from women with preeclampsia: Plasma collected from women who developed preeclampsia during pregnancy will be analyzed for mechanism of NETs formation.
- Plasma from women with normal pregnancies: Plasma collected from women with normal pregnancies will be analyzed for mechanism of NETs formation.

SUMMARY:
Formation of neutrophil extracellular traps (NETs) is a process of activation of neutrophils, which then generate filaments containing DNA, enzymes and extracellular histones. Two mechanisms of formation of NETs are described in the literature: vital mechanism via Toll Like Receptors (TLRs) and suicidal mechanism, dependent on the reactive oxygen species (ROS) pathway. The description of these two mechanisms of formation of NETs is recent and no data exist in the context of pregnancy.

DETAILED DESCRIPTION:
This is a descriptive pilot study on a ready-constituted biobank. It is an ancillary study to a previous cohort (RCB number: 2014-A01120-47, NCT01736826).

Pregnancy generates an increased risk of thrombosis, and placenta-mediated diseases constitute a risk factor for cardiovascular pathologies responsible for significant maternal-fetal morbidity and mortality. Understanding and exploring the cellular and molecular mechanisms of dysfunctions of the vascular-placental interface could provide arguments to understand the systemic vascular risk, characterize it and finally detect it on the basis of new markers, thus opening the way for targeted preventive management to reinforce the general principles of precision medicine.

Formation of NETs is a process of activation of neutrophils, which then generate filaments containing DNA, enzymes and extracellular histones. Formation of NETs occurs in pregnancy and is increased in vascular-placental complications. It can be studied by measuring circulating histones, particularly the citrullinated histone H3. Levels of this modified histone H3, as well as those of two other modifications, have recently been shown to increase during pregnancy. These levels have also been shown to be even greater in pregnancy complications.

Furthermore, two mechanisms of formation of NETs are described in the literature: vital mechanism via Toll Like Receptors (TLRs) and suicidal mechanism, dependent on the reactive oxygen species (ROS) pathway. The description of these two mechanisms of formation of NETs is recent and no data exist in the context of pregnancy.

The aim of this study is to describe the part of these two mechanisms in normal and complicated pre-eclampsia pregnancies in order to obtain a better physiopathological knowledge of pre-eclampsia to propose new circulating biomarkers and to develop new therapeutic strategies for placental vascular pathologies.

ELIGIBILITY:
Not applicable as this study is on samples from a biobank.

Inclusion criteria:

The inclusion criteria for the previous cohort (NCT01736826) were:

* pregnant women followed at Nimes University hospital for normal pregnancy or pregnancy with placental vascular pathology (pre-eclampsia and/or intra-uterine growth retardation).
* The patient must have given her free and informed consent and signed the consent form.
* The patient must be a member or beneficiary of a health insurance plan
* Only women are included
* Patients are at least 18 years old

Exclusion Criteria:

Not applicable as this is a study on samples from a biobank. The non-inclusion criteria of the previous cohort (NCT01736826) were :

• twin pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: The study is based on frozen plasma samples from pregnant women, taken at the time of them giving birth from among the 85 women who constituted the previous cohort (NCT01736826). Thirteen of these women had had normal pregnancies and thirteen had developed pre-eclampsia. Cases are matched on maternal age, clinical event (delivery) and gestational age will be included from the previous cohort (NCT01736826).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate vital mechanism of NETs formation between pregnant women with normal pregnancies and those developing preeclampsia. | 3 months
  Evaluation of vital mechanism of NETs formation between pregnant women with normal pregnancies and those developing preeclampsia.

SECONDARY OUTCOMES:
To compare the proportion of vital mechanism of NETs formation in the presence or absence of a TLR-blocking antibody within each group: normal pregnancy and preeclamptic pregnancy. | 3 months
  Evaluation of the proportion of vital mechanism of NETs formation in the presence or absence of a TLR-blocking antibody within each group: normal pregnancy and preeclamptic pregnancy.
To compare the proportion of vital mechanism of NETs formation in the presence of a TLR-blocking antibody between pregnant women with normal pregnancies and those developing preeclampsia. | 3 months
  Evaluation of the proportion of vital mechanism of NETs formation in the presence of a TLR-blocking antibody between pregnant women with normal pregnancies and those developing preeclampsia.
To compare vital and suicidal mechanisms of NETs formation between pregnant women with a normal pregnancy and those developing preeclampsia. | 3 months
  Evaluation of vital and suicidal mechanisms of NETs formation between pregnant women with a normal pregnancy and those developing preeclampsia.
To compare vital and suicidal mechanisms of NETs formation in the presence or absence of a TLR blocking antibody or ROS inhibitor (DPI) separately within each group: normal pregnancy and preeclamptic pregnancy. | 3 months
  Evaluation of vital and suicidal mechanisms of NETs formation in the presence or absence of a TLR blocking antibody or ROS inhibitor (DPI) separately within each group: normal pregnancy and preeclamptic pregnancy.
To compare vital and suicidal mechanisms of NETs formation in the presence of TLR blocking antibody or ROS inhibitor (DPI) between pregnant women with normal pregnancy and those developing preeclampsia. | 3 months
  Evaluation of vital and suicidal mechanisms of NETs formation in the presence of TLR blocking antibody or ROS inhibitor (DPI) between pregnant women with normal pregnancy and those developing preeclampsia.
To compare the proportion of suicidal mechanism of NETs formation between pregnant women with a normal pregnancy and those developing preeclampsia. | 3 months
  Evaluation of the proportion of suicidal mechanism of NETs formation between pregnant women with a normal pregnancy and those developing preeclampsia.
To compare suicidal mechanism of NETs formation in the presence or absence of ROS inhibitor (PGD) separately within each group: normal pregnancy and preeclamptic pregnancy. | 3 months
  Evaluation of suicidal mechanism of NETs formation in the presence or absence of ROS inhibitor (PGD) separately within each group: normal pregnancy and preeclamptic pregnancy.
To compare the proportion of suicidal mechanism of NETs formation in the presence of an ROS inhibitor (PGD) between pregnant women with a normal pregnancy and those developing preeclampsia. | 3 months
  Evaluation of the proportion of suicidal mechanism of NETs formation in the presence of an ROS inhibitor (PGD) between pregnant women with a normal pregnancy and those developing preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Chair — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Guillotin F, Fortier M, Portes M, Demattei C, Mousty E, Nouvellon E, Mercier E, Chea M, Letouzey V, Gris JC, Bouvier S. Vital NETosis vs. suicidal NETosis during normal pregnancy and preeclampsia. Front Cell Dev Biol. 2023 Jan 5;10:1099038. doi: 10.3389/fcell.2022.1099038. eCollection 2022. PMID 36684420